CLINICAL TRIAL: NCT01493453
Title: A Phase I Study of Adoptive Transfer of Autologous Tumour Antigen-Specific T Cells With Pre-conditioning Chemotherapy and Intravenous IL2 in Patients With CD19 Positive Malignancy
Brief Title: A Phase I Study of CD19 Specific T Cells in CD19 Positive Malignancy
Acronym: CD19
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Investigation into serious breach
Sponsor: The Christie NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05_DOG05_18
Record Dates: First submitted 2011-12-14; First posted 2011-12-16 (Estimated); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: CD19 Positive Non-Hodgkin Lymphoma
MeSH Terms: interventions — Interleukin-2; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm - aCD19z cells, interleukin 2, Chemotherapy (Experimental)
  Interventions: Genetic: aCD19z cells, IL2, pre conditioning Cyclophosphamide & Fludarabine

INTERVENTIONS:
Genetic: aCD19z cells, IL2, pre conditioning Cyclophosphamide & Fludarabine — aCD19z T cells IV Day 1. The dose of aCD19z T cells will be determined by dose escalation scheme, starting at 10*9 IL2 given as 15 minute IV infusion every eight hours for up to 12 doses Cyclophosphamide (C) 15mg/kg day -7 and day -6, Fludarabine (F) 25mg/m2 day -5 to day -1.

SUMMARY:
In particular circumstances T cells can be an effective treatment for malignant disease, for example, donor lymphocyte infusions following allogeneic transplants or treatment of EBV related lymphomas post allograft. However, many common cancers are poorly recognised by the immune system in part because of a lack of suitable T cell targets and in part because of defects in antigen presentation by tumours (Garrido, et al 1997). Genetically modified T cells engineered to express chimeric immune receptors (CIRs) on their cell surface can bypass the need for MHC presentation and thus represent an attractive approach to immunotherapy (Gross, et al 1989).

DETAILED DESCRIPTION:
CD19 is an Immunoglobulin-like 95kDa glycoprotein that is expressed on all B lymphocytes until differentiation into terminal effector cells (Tedder and Isaacs 1989). It plays an important role in regulating cell signalling thresholds and also as a costimulatory molecule for B cell receptor signalling (Tedder, et al 1997). CD19 is present on the majority of B-CLL, B-ALL, and both low and high grade non-Hodgkin lymphomas (NHL). It is rarely lost during the process of neoplastic transformation and is not expressed on haematopoetic stem cells. B cell malignancies are often highly responsive to chemotherapy, with cures possible in significant numbers of those with high grade tumours. However, improved treatments are needed for those with low grade tumours and those with high grade tumours who relapse after conventional therapy.

In recent years the introduction of Rituximab, a CD20 monoclonal antibody, into clinical practice has increased the options available for the treatment of NHL (Maloney, et al 1994). The success of Rituximab and other monoclonal antibodies has demonstrated that B cell malignancies may be particularly suitable as a target for immunotherapy. However, there are number of potential advantages of T cells engineered to express a CIR over monoclonal antibody therapies. Firstly, the possibility of in vivo T cell persistence and expansion may enable stable expression of the CIR over a prolonged period of time (Walker, et al 2000). Secondly, homing to the tumour site may mean that T cells need not rely on diffusion to achieve localisation (Balkwill 2004, Mitsuyasu, et al 2000) and thirdly following tumour recognition T cells can produce cytokines that may recruit and activate other effector cells. An alternative to CIR engineered T cells is the generation of peptide specific T cells. Lymphoma models suggest these can be effective (Armstrong, et al 2002, Armstrong, et al 2004), but to produce clinically applicable numbers of T cells is technically demanding and there is a lack of generic peptide target antigens in lymphoma.

One potential problem in the use of CIR engineered T cells in general is that tumour associated antigens are frequently expressed at low levels on normal tissues, thus providing the potential for autoimmunity. Targeting B cell malignancies with CD19 specific T cells is attractive because whilst CD19 is expressed on B cells and the majority of B cell malignancies it is not expressed on any other cell type. It is clear from clinical use of anti-CD20 antibodies that prolonged depletion of B cells (>6 months) is safe (Plosker and Figgitt 2003) and that even in patients with hereditary B cell deficiency immunoglobulin infusion restores normal health in most patients (Ochs and Smith 1996).

The Investigators have therefore propose a clinical trial using T cells expressing a CD19 targeting CIR by retroviral transduction of the CIR into activated T cells in order to target B cell malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed CD19 positive non-Hodgkin Lymphoma with evidence of persistent or progressive disease and poor prognosis as discussed in detail in section 1.5
* Written informed consent and the ability of the patient to co-operate with study treatment, procedures and follow up must be ensured and documented.
* Age equal to or greater than 18 years.
* World Health Organisation (WHO) performance status of 0 or 1 (appendix 1).
* Life expectancy >3months.
* LVEF > 50% as measured by MUGA scan
* Haematological and biochemical indices:

Haemoglobin (Hb)≥ 10.0 g/dl neutrophils ≥ 1.0 x 109/L platelets (Plts)≥ 100 x 109/L

Any of the following abnormal baseline liver function tests:

serum bilirubin ≤ 1.5 x upper limit of normal (ULN) alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) and /or alkaline phosphatase (ALP)≤ 5 x ULN Serum creatinine ≤ 0.14 mmol/L

* Female patients of child-bearing potential are eligible, provided they have a negative serum or urine pregnancy test prior to enrolment and agree to use appropriate medically approved contraceptive precautions for four weeks prior to entering the trial, during the trial, and for six months afterwards.
* Male patients must agree to use barrier method contraception during the trial and for six months afterwards.
* Measurable disease as defined by RECIST criteria (appendix 3).

Exclusion Criteria:

* Radiotherapy, biological therapy, endocrine therapy, immunotherapy, systemic steroids, or chemotherapy during the previous four weeks (six weeks for nitrosoureas and Mitomycin-C) prior to treatment or during the course of the trial.
* All toxic manifestations of previous treatment must have resolved. Exceptions to this are alopecia or certain Grade 1 toxicities which in the opinion of the Investigator and Trial Sponsor should not exclude the patient.
* Participation in any other clinical trial within the previous 30 days or during the course of this trial.
* Previous participation in a Gene Therapy trial.
* Previous allogeneic transplant.
* Patients who are high medical risks because of non-malignant systemic disease, including those with active infection, uncontrolled cardiac or respiratory disease, or other serious medical or psychiatric disorders which in the Investigator's opinion would not make the patient a good candidate for the clinical trial.
* Concurrent serious infections within the 28 days prior to entry to the trial.
* Current malignancies at other sites, with the exception of adequately treated cone-biopsied in situ carcinoma of the cervix uteri and basal or squamous cell carcinoma of the skin.
* Patients known or found to be serologically positive for Hepatitis B, C, HIV or HTLV.
* History of autoimmune disease.
* Evidence of CNS involvement.
* Patients who are likely to require systemic steroids or other immunosuppressive therapy.
* Pregnant and lactating women.
* Radiotherapy to >25% skeleton.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2008-03; Primary Completion 2014-12 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
To asses aCD19z T cell survival and aCD19z T cell toxicity in patients, & The dose of aCD19z T cells required to give optimal survival of these cells in the circulation | Week 6

SECONDARY OUTCOMES:
To assess whether aCD19z T cells in the circulation are functional | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- The Christie NHS Foundation Trust, Manchester, United Kingdom